CLINICAL TRIAL: NCT03024515
Title: A Pilot Randomized Open-labeled Study Comparing a Structured Titration Method of immediate-and Sustained- Release Oxycodone Versus Opioids Titration of Investigators' Choice in Advanced Cancer Patients in Hong Kong
Brief Title: Opioids Titration Study in Advanced Cancer Patients in Hong Kong
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, CCTU, Assistant Professor (Clinical), Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYM012
Record Dates: First submitted 2016-11-23; First posted 2017-01-19 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Pain Control
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Practice Arm (Experimental): Standard Practice Arm with opioids titration of physicians' choice
  Interventions: Drug: opioids titration
- Structured Tritration Arm (Experimental): Structured titration method with predefined titration steps with the use of oxycodone immediate-release and oxycodone sustained-release preparations.
  Interventions: Drug: predefined titration steps

INTERVENTIONS:
Drug: opioids titration — Standard Practice Arm
  Arms: Standard Practice Arm
Drug: predefined titration steps — comprising of oxycodone immediate release (OXYNORM) and oxycodone sustained release (OXYCONTIN) in pre-defined doses and frequencies
  Arms: Structured Tritration Arm

SUMMARY:
Pain is a common symptom that is experienced by patients with advanced cancer. Whilst mild pain can usually be controlled with simple analgesics, more severe pain may require initiation of opioid analgesics. The World Health Organization (WHO) has developed a specific guideline for titration of analgesics. Known as the WHO Pain Ladder, patients who have severe pain despite non-opioid and weak opioid analgesics are advised to step up to level 3 - "Strong Opioids". Morphine is the most common opioid strong analgesic prescribed in Hong Kong. To the best of our knowledge, there is no formal opioid pain control guideline developed for cancer patients in Hong Kong. The prescription practices of various physicians who treat advance cancer patients, including oncologists and palliative care physicians have never been audited or standardized.

Furthermore, there are inherent issues with the administration of oral morphine. Currently, only one fixed concentration is available in a liquid formulation. Patients are known to have difficulties in receiving the appropriate dose. Accurate measurement of the volume required is extremely difficult, and many a times patients will report to have spilled the oral morphine during decanting, or will report that they have not been taking adequate doses because they are worried that they will decant too much into a spoon or syringe and overdose themselves.

Oxycodone is a semisynthetic strong opioid analgesic, which has recently been introduced to Hong Kong. It is formulated as a capsule, and again, 2 preparations (sustained-release (Oxycontin) and immediate release (Oxycodone IR)) are available. Inherent advantages include ease of administration; different groups have previously reported less adverse effects and better treatment compliance. However, to date, there has been no prospective 'head-to-head' comparison have ever been carried out comparing this with the traditional, well-accepted methods.

The purpose of this study is to assess whether or not the use of Oxycontin and Oxycodone IR may be superior to traditional medication choices and schedules in terms of time required for onset of pain control, the side effect profile, patients' tolerability and compliance to treatment. Interestingly, through this randomized open-label prospective study, we also aim to capture information on current opioid prescription practices by clinicians who manage patients with advanced cancers, which will be useful for us to consider the establishment of territory-wide treatment guidelines at a later juncture.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient with moderate to severe cancer pain, and:
2. Opioid naïve patients, who were administrated NSAIDs or weak opioids and currently with poor pain control, intend to be treated with strong opioids
3. For the patients who need long term administration of hormone or targeting therapy or bisphosphonates therapy, the treatments will maintain from 3 days prior to randomization to end of the study as much as possible.
4. For patients who need radiotherapy or chemotherapy, these therapies should be conducted during maintaining phase and completed as assuring as possible before last follow-up.

Exclusion Criteria:

1. The pure neuropathic pain or unexplained pain, pain that only occurs during moving; Acute pain
2. The patients who are not applicable for oral administration
3. Any disease that may lead to respiration inhibition of the subjects
4. Monoamine oxidase inhibitor (MAOI) was administrated one week before randomization;
5. There are abnormal results, with obvious clinical significance, from lab testing, such as the creatinine is ≥2-fold of upper limit of normal value, or ALT or AST is ≥2-fold of upper limit of normal value, or liver function is Child C grade;
6. There are potential gastrointestinal diseases or the risk of surgical operation, which may lead to gastrointestinal stenosis, blind loop or gastrointestinal obstruction;
7. Patients have been exposed to prolonged-release oxycodone tablets or other strong opioids drugs before study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-08-23 (Actual); Primary Completion 2020-12-07 (Actual); Study Completion 2020-12-07 (Actual)

PRIMARY OUTCOMES:
Time to stabilization of pain control during titration phase | 1 year

SECONDARY OUTCOMES:
Time of analgesic onset | 1 year
Number of breakthrough medications required during the titration phase | 1 year
Quality of Life assessments using the EORTC QLQ-C15-PAL instrument | 1 year
A descriptive assessment of opioids prescription practice amongst practicing oncologists in Hong Kong | 1 year
Safety profile and adverse events | 1 year
Descriptive summary of the use of opioids and titration by practicing clinicians | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Oncology, Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No